CLINICAL TRIAL: NCT04058795
Title: Using a SMART Design to Optimize PTSD Symptom Management Strategies Among Cancer Survivors
Brief Title: PTSD Mobile App for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00103154
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-04

CONDITIONS: Posttraumatic Stress Disorder; Cancer
Keywords: PTSD; Depression; Anxiety; Distress; Digital Health; mHealth
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Neoplasms; Depression; Anxiety Disorders | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cancer Distress Coach (CaDC) (Experimental): Participants in this group will get the mHealth CaDC app, which will give them tools based on cognitive behavioral therapy principles to manage their stress.
  Interventions: Behavioral: Cancer Distress Coach (CaDC) App
- CaDC and mCoaching (Experimental): Participants in this group will get both the CaDC app and weekly clinician support.
  Interventions: Behavioral: CaDC + mCoaching
- mCBT (Experimental): Participants in this group will get 8-sessions with a therapist to receive cognitive behavioral therapy (CBT).
  Interventions: Behavioral: mCBT
- Control (No Intervention): Participants in this group can use mental health services commonly available to all cancer patients at their local medical facility but will not receive access to the CaDC app.

INTERVENTIONS:
Behavioral: Cancer Distress Coach (CaDC) App — an app that provides participants with tools to manage their stress in the moment they experience it.
  Arms: Cancer Distress Coach (CaDC)
Behavioral: CaDC + mCoaching — The CaDC app plus weekly clinician support which provides support in navigating the app, encouraging adherence to the use of the CaDC, and providing guidance in choosing treatment strategies.
  Arms: CaDC and mCoaching
Behavioral: mCBT — 8 mobile sessions with a therapist to receive cognitive behavioral therapy.
  Arms: mCBT

SUMMARY:
The purpose of this study is to use a stepped-care approach in treating symptoms of posttraumatic stress disorder (PTSD). The information learned by doing this study may help us to develop some target treatments for PTSD symptoms in survivors of stem cell transplant.

Participants in this study will be randomized to a mobile app or usual care. An assessment will be made after 4 weeks and a determination made of adding more intensive treatment. Participants will be asked to complete a questionnaire 4 times over a period of 6 months, at the time your participation is complete.

ELIGIBILITY:
Inclusion Criteria:

* Completion of autologous or allogeneic HCT 1-5 years previously
* Partial or complete remission (NED), may be receiving chemoprevention
* Absence of severe psychological impairment (eg hospitalization for suicidality)
* Approved for contact by oncologist
* Able and willing to participate in a one-hour baseline interview
* No prior CBT for PTSD
* Owns a smart device with internet and email access
* Able to read and write English
* Significant PTSD symptoms as indicated by at least one of the following two criteria: probable cancer-related PTSD on the PCL5 by using the symptom cluster criteria; subthreshold or partial PTSD symptoms as determined by endorsement of reexperiencing cluster and less than or equal to 1 other symptom cluster

Exclusion Criteria:

* If the participant does not fulfill the inclusion criteria

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2021-01-24 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptoms measured by the PTSD checklist (PCL5) | baseline, 4 weeks, 12 weeks
  PCL5 is 20 item instrument scored 0-4, with 0 being "Not at all" and 4 being "Extremely"

SECONDARY OUTCOMES:
Change in distress measured by the Distress Thermometer v. 2018 | baseline, 4 weeks, 12 weeks, and 6 months
  Distress Thermometer v. 2018 is a one item instrument scored 0-10, with 0 being "No distress" and 10 being "Extreme distress"
Change in PTSD symptoms measured by the PTSD checklist (PCL5) | baseline, 12 weeks, 6 months
  PCL5 is 20 item instrument scored 0-4, with 0 being "Not at all" and 4 being "Extremely"
Change in Quality of Life measured by the PROMIS QOL | baseline, 4 weeks, 12 weeks, and 6 months
  PROMIS QOL is a 10 item instrument scored 1-5, with 1 being "Never" and 5 being "Always"
Change in depression as measured by the PROMIS | baseline, 4 weeks, 12 weeks, and 6 months
  PROMIS is an 8 item instrument scored 1-5, with 1 being "Never" and 5 being "Always"
Change in anxiety as measured by the PROMIS | baseline, 4 weeks, 12 weeks, and 6 months
  PROMIS is an 8 item instrument scored 1-5, with 1 being "Never" and 5 being "Always"
Change in self-efficacy as measured by the Self-efficacy for Chronic Disease | baseline, 4 weeks, 12 weeks, and 6 months
  Self-efficacy for Chronic Disease is a 6 item instrument scored 1-10, with 1 being "Not at all confident" and 10 being "totally confident"
User satisfaction as measured by a survey | baseline, 4 weeks, 12 weeks, and 6 months
  Team developed survey that will include questions regarding the participant's experience

CONTACTS AND LOCATIONS:
Overall Officials: Sophia K Smith, PhD, MSW, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Memorial Sloan Kettering, New York, New York
  - Duke University, Durham, North Carolina
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith SK, Manschot C, Kuhn E, Laber E, Somers TJ, Syrjala KL, Applebaum AJ. Assessing the utility of the PC-PTSD-5 as a screening tool among a cancer survivor sample. Cancer. 2024 Dec 1;130(23):4118-4126. doi: 10.1002/cncr.35504. Epub 2024 Aug 14. PMID 39141666
- See also: Study Website — https://sites.duke.edu/transplantsurvivorcoach/contact-us/

DOCUMENTS (1):
  • Informed Consent Form (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT04058795/ICF_000.pdf